CLINICAL TRIAL: NCT07217275
Title: Rise With Resilience: A Clinical Trial Examining Mindfulness Training for Enhancing Recovery in Injured Student-Athletes
Brief Title: Rise With Resilience
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Collegiate Athletic Association - NCAA (Unknown)
Responsible Party: Principal Investigator, Nicholas A. Giordano, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025P011851
Record Dates: First submitted 2025-10-13; First posted 2025-10-15 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Athletic Injuries; Sport Injuries
Keywords: Orthopedic surgery; Student Athletes; Mindfulness skills
MeSH Terms: conditions — Athletic Injuries | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Resiliency Model (CRM) (Experimental): Athletes randomized to the intervention will receive education before surgery. The intervention includes pairing participants with a specialist who will introduce mindfulness skills to athletes, educate them on how to apply the skills, and observe athletes practicing the skills via Zoom®.
  Interventions: Other: Community Resiliency Model (CRM)
- Standard of Care (SOC) (Active Comparator): Athletes randomized to the control group will receive standard of care, written instructions, and handouts on postoperative pain management interventions.
  Interventions: Other: Control

INTERVENTIONS:
Other: Community Resiliency Model (CRM) — CRM is an evidence-based mindfulness approach that provides patients with a biological perspective on behavioral health and stress reactions. CRM teaches six (6) mindfulness-based skills to address body sensation perception to attenuate symptoms of stress and anxiety, which in turn contribute to reducing pain and stress response. Trained specialists will introduce mindfulness skills to athletes, educate them on how to apply the skills, and observe athletes practicing the skills via Zoom®. Participants will be randomized to work with a mindfulness specialist at the baseline visit for 90 minutes and at follow-up visits for 15-30 minutes over Zoom®. The team's mindfulness specialists will deliver the evidence-based mindfulness training.
  Other Names: Virtual Intervention
  Arms: Community Resiliency Model (CRM)
Other: Control — Participants will receive written discharge instructions on postoperative pain management interventions given to all patients seeking care at Emory. The handout includes guidance on when to take prescribed pain medications and how to implement non-pharmacological pain management approaches, such as cryotherapy or aroma therapy. To mitigate attention biases, study staff and clinical staff will meet with control arm participants at each follow-up visit for 15-30 minutes to review the handout. This minimally enhanced usual care attention-based control group design has been successfully utilized in other trials to mitigate biases and dropouts.
  Other Names: Standard of Care (SOC)
  Arms: Standard of Care (SOC)

SUMMARY:
The objective of this study is to investigate differences in postoperative pain, physical health, and mental health outcomes between participants receiving evidence-based mindfulness training and those who do not.

Over 200,000 injuries are estimated to occur among National Collegiate Athletic Association (NCAA) athletes annually. For many, these injuries can be season-ending, exacerbating physical, mental, and social well-being. Student-athletes face distinctive challenges compared to traditional students, such as balancing academic and athletic demands, pressures to perform well on and off the field, and the physical demands of competition, all of which can lead to worse mental and emotional outcomes if not properly managed. Injuries heighten stress levels among athletes, remove them from competition, and force students to integrate treatment regimens into already packed academic schedules.

DETAILED DESCRIPTION:
In this study, researchers will investigate how student-athletes can enhance their recovery following surgery for an injury by incorporating mindfulness-based practices.

Athletic performance, physical output, and overall wellness have been shown to improve when athletes incorporate evidence-based mindfulness and cognitive skills. Yet, minimal research has examined how cognitive and mindfulness skills can be leveraged specifically by injured student athletes to facilitate return to play, mitigate stress, and support academic performance following surgery. This randomized clinical trial will recruit college athletes undergoing surgery due to injury and randomize them to work with an expert on implementing skills from the Community Resiliency Model® (CRM).

Over the span of three months after surgery, the interdisciplinary research team will compare patient-reported outcomes and objective recovery measures from wrist-worn actigraphy devices to determine the impact of educating athletes on incorporating CRM skills that enhance well-being following surgery, compared to standard of care (SOC) written discharge instructions. Participants will complete questionnaires in person and/or via email about their general health and their pain at each appointment.

ELIGIBILITY:
Inclusion Criteria:

* College student athletes 18-26 years old,
* Scheduled for orthopedic surgery due to sports medicine injuries (e.g., anterior cruciate ligament tears, meniscus injury, rotator cuff injury, etc.)

Exclusion Criteria:

* Individuals unable to provide consent
* Undergoing revision procedures
* Individuals without access to an internet-connected device.
* Unable to speak English

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function | Baseline (pre-surgery), 2 weeks, 6 weeks, and 3 months (post-surgery)
  PROMIS Physical Function measures participants' self-reported capability to conduct physical activity. This includes capturing function in upper extremities and lower extremities (walking or mobility) as well as a respondent's ability to conduct activities of daily living. There are 4-items on the short form questionnaire and respondents report their capabilities to perform each task on a Likert scale from 5, "without any difficulty", to 1, "unable to do". All 4-items' saw scores are summed before being transformed into t-scores ranging from 0 to 100. Higher scores are better and indicate greater physical function.
Opioid utilization | Baseline (pre-surgery), 2 weeks, 6 weeks, and 3 months (post-surgery)
  Inpatient and operating room opioid utilization will be extracted from the electronic health record (EHR) by study staff upon participants' discharge from the hospital. Opioid medication dosage will be transformed to a total universal measure known as morphine milligram equivalent (MME). MME will be averaged over the length-of-stay (LOS) for a daily dosage, known as MME/day. Additionally, the study team will review the participants' EHR at each study time point up to 3 months to determine MME throughout postoperative recovery and rehabilitation. Higher values indicate a greater dosage per day.
Pain numerical rating scale (NRS) | Baseline (pre-surgery), 2 weeks, 6 weeks, and 3 months (post-surgery)
  The NRS requires respondents to rate the intensity of their pain on a defined scale from 0, "no pain", to 10, 'the worst pain imaginable". The NRS is a commonly used pain assessment tool in both clinical practice and research. Higher scores indicate worse pain.

SECONDARY OUTCOMES:
Mindful Attention Awareness Scale (MAAS) | Baseline (pre-surgery), 2 weeks, 6 weeks, and 3 months (post-surgery)
  The MAAS is a validated 15-item scale designed to assess a core characteristic of dispositional mindfulness, namely, open or receptive awareness of and attention to what is taking place in the present. Each item is rated on a 6-point Likert scale (1 = Almost Always, 6 = Almost Never). The mean or total score is calculated, with higher scores indicating greater mindfulness (i.e., more awareness and attention to the present moment), and lower scores indicating more automatic or distracted behavior.
Connor-Davidson Resilience Scale (CD-RISC) | Baseline (pre-surgery), 2 weeks, 6 weeks, and 3 months (post-surgery)
  The Connor-Davidson (CD) Resilience Scale (RISC) assesses the ability to recover from a stressful event. The abbreviated version of this scale, CD-RISC-2, uses two questions from the original CD-RISC that capture the essence of resilience. Question 1, which asks if the respondent is "Able to adapt to change," and question 8, which asks the respondent whether they "Tend to bounce back after illness or hardship," are used in this 2-item abbreviated measure. Range: 0-8 (Each item scored 0 = not true at all to 4 = true nearly all the time.)The abbreviated nature of this scale allows for a quick, valid, and reliable measure of a respondent's self-perceived resilience in the face of a potentially stressful event such as orthopedic surgery. Scoring: Sum the two items. Higher scores = greater resilience. Example: 0-2 = very low resilience; 7-8 = very high resilience.
Injury-Psychological Readiness to Return to Sport scale (I-PRRS) | Baseline (pre-surgery), 2 weeks, 6 weeks, and 3 months (post-surgery)
  This 10-item scale is used to assess mental readiness, asking questions about confidence to play, ability to give 100% effort, and confidence in the ability to be successful upon return to play. Response format: 0-10 Likert scale 90 = Not at all confident/ready and 10 = Very confident/completely ready). Each item asks how confident the athlete feels about aspects such as: Performing at their pre-injury level, coping with pain, re-injury fears, trust in the injured body part, and overall readiness to return. Scoring range: 0-100, with higher scores indicating greater psychological readiness to return to sport and lower scores = more anxiety, doubt, or lack of confidence
Resilience Scale for Adults | Baseline (pre-surgery), 2 weeks, 6 weeks, and 3 months (post-surgery)
  This 33-item scale aims to characterize a respondent's resilience in several contexts and provides a scale ranging from extremely positive outlooks to extremely negative. For example, in response to being asked "in difficult times, my family…", a scale ranging from "keeps a positive outlook on the future" to "views the future as gloomy" is provided to respondents. The breadth of question types included in this resilience scale makes it a comprehensive evaluation of an athlete's ability to respond in times of struggle. Range: 33-231, with each item scored 1-7. Scoring: Mean or total score. Higher scores indicate a greater resilience (stronger protective factors and adaptability), and lower scores indicate lower resilience or more vulnerability to stress.
ACL-Return to Sport after Injury (ACL-RSI) scale | Baseline (pre-surgery), 2 weeks, 6 weeks, and 3 months (post-surgery)
  This 12-item questionnaire asks questions regarding an athlete's emotions, confidence in performance, and appraisal of risk specifically related to knee injury. While this scale has been used exclusively for evaluation of an athlete's return to sport in response to knee injury, it has application to all orthopedic related sports injuries that require surgical intervention. Some questions include: Are you nervous about playing your sport? Do you feel relaxed about playing your sport? Are you afraid of accidentally injuring your knee by playing your sport? Are you confident that you can perform at your previous level of sport participation? Do thoughts of having to go through surgery and rehabilitation again prevent you from playing your sport? Scoring extremely low demonstrates significantly worse return to play outcomes.
Actigraphy based sleep data | Baseline (pre-surgery) and 2 weeks (post-surgery)
  The sleep data will be computed using the Cole-Kripke algorithm, which accurately distinguishes sleep from wakefulness approximately 88% of the time. Participants will receive a screenless actigraphy device and will be trained on how to wear it on their wrist. Higher sleep values indicate better or longer sleep.
Actigraphy based physical activity intensity | Baseline (pre-surgery) and 2 weeks (post-surgery)
  Physical activity intensity will be captured using wrist actigraphy. Participants will receive a screenless actigraphy device and will be trained on how to wear it on their wrist. More frequent periods of higher intensity indicate improved activity.
Actigraphy based activity time | Baseline (pre-surgery) and 2 weeks (post-surgery)
  Activity time will be captured using wrist actigraphy. Participants will receive a screenless actigraphy device and will be trained on how to wear it on their wrist. Longer duration indicates more time spent actively.
Actigraphy based activity (steps) | Baseline (pre-surgery) and 2 weeks (post-surgery)
  Steps will be captured using wrist actigraphy. Participants will receive a screenless actigraphy device and will be trained on how to wear it on their wrist. More steps per day indicate greater physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A Giordano, PhD, RN, Principal Investigator — Emory University
Locations (1):
- Emory Orthopaedics and Spine Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No